CLINICAL TRIAL: NCT05776771
Title: The Spine Phenome Project: Enabling Technology for Personalized Medicine
Brief Title: The Spine Phenome Project
Status: Recruiting | Type: Observational
Sponsor: Ohio State University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Principal Investigator, William Marras, Director of SRI, Ohio State University
Other Study IDs: 2020H0250; 4UH3AR076729-02 (NIH)
Record Dates: First submitted 2023-02-06; First posted 2023-03-20 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2024-05

CONDITIONS: Low Back Pain; Neck Pain
MeSH Terms: conditions — Low Back Pain; Neck Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Low Back Pain: Subjects with Low Back Pain
- Neck Pain: Subjects with Neck Pain
- Control/Insincere: Subjects with healthy spines, who have no neck or low back pain

SUMMARY:
The goal of this observational trial is to compare the health history and motion capabilities of participants with low back pain disorders to participants with healthy spines. The main question[s] it aims to answer are to:

1. Primary outcomes of this research effort include composite measures that differentiate between control and patient populations, predict injury or reinjury risk, identify low back and neck pain patient phenotypes, and evaluate treatment effectiveness.
2. Secondary outcomes of this research effort include an assessment of wearable motion sensor accuracy, characterization of motion assessment utility, biopsychosocial profiling of control and low back and neck pain patient populations, and differentiation of sincere and insincere motion assessment efforts.

Participants will complete questionnaires and wear a motion monitor that will assess your back and/or neck. This session will be approximately 40-70 minutes. The research team will follow up with participants at 3 month, 6 months, 1 year, 2 years, 5 years to complete a short series of questionnaires and a motion assessment test.

ELIGIBILITY:
Controls/Insincere

Inclusion Criteria

* Age 18 and older
* Able to stand for 20 minutes
* Able to speak, read, and understand English

Exclusion criteria:

* Known pregnancy
* Currently seeing or planning to see a medical provider for low back or neck pain
* History of chronic low back or neck pain lasting longer than 3 months
* Blind or severe uncorrected vision problems that prevent participant from reading a tablet or laptop screen
* Deaf or hearing problems that prevent the participant from hearing verbal instructions
* Actively being treated by a medical provider for concussion
* Known severe spinal deformity requiring medical treatment (e.g. scoliosis)
* Has been diagnosed by a medical provider with severe vertigo, fainting, narcolepsy, or balance disorders with high risk for falling
* Any known fractures within the last 3 months that will interfere with the motion assessment
* History of spine fracture
* Current condition requiring immobilization or bracing of the spine
* History of spine surgery (e.g. fusion, micro-discectomy, or artificial disc replacement)
* History of brain or spine cancer
* Currently or within the last 90 days, been treated for cancer with chemotherapy or radiation therapy
* Known severe osteoporosis requiring medical treatment and physician-recommended physical restrictions
* Current open wounds or medical device entry points where the harnesses will be placed on the neck, back, or hips
* Current osteomyelitis or spine infection
* Any other reason that a treating physician, researcher, or participant determines it is unsafe for a patient to perform test

Low Back Pain Patients

Inclusion Criteria

* Age 18 and older
* Currently seeking medical consult with primary complaint of low back pain
* Able to speak, read, and understand English
* Able to stand for 10 minutes

Exclusion criteria:

* Known pregnancy
* Blind or severe uncorrected vision problems that prevent participant from reading a tablet or laptop screen
* Deaf or hearing problems that prevent the participant from hearing verbal instructions
* Current low back pain is the result of a traumatic injury (wreck, fall, etc.) that occurred within the last 3 months OR is positive for spine instability with imaging
* Has spinal fusion across 4 or more lumbar disc levels.
* Actively being treated by a medical provider for concussion
* Known severe spinal deformity requiring medical treatment (e.g. scoliosis)
* Has been diagnosed by a medical provider with severe vertigo, fainting, narcolepsy, or balance disorders with high risk for falling
* Any known fractures within the last 3 months that will interfere with the motion assessment
* Any known spine fractures within the last 6 months
* Known unstable spondylolisthesis (i.e. standing 3mm of movement on flexion/extension film)
* Current condition requiring immobilization of the spine
* History of brain or spine cancer
* Currently or within the last 90 days, been treated for any cancer with chemotherapy or radiation therapy
* Known severe osteoporosis requiring medical treatment and physician-recommended physical restrictions
* Current open wounds or medical device entry points where the harnesses will be placed on the back or hips
* Current osteomyelitis or spine infection
* Any other reason that a treating physician, researcher, or participant determines it is unsafe for a patient to perform test

Neck Pain Patients

Inclusion Criteria

* Age 18 and older
* Currently seeking medical consult with primary complaint of neck pain
* Able to speak, read, and understand English
* Able to stand for 10 minutes

Exclusion criteria:

* Known pregnancy
* Blind or severe uncorrected vision problems that prevent participant from reading a tablet or laptop screen
* Deaf or hearing problems that prevent the participant from hearing verbal instructions
* Current neck pain is the result of a traumatic injury (wreck, fall, etc.) that occurred within the last 3 months OR is positive for spine instability with imaging
* Has spinal fusion across 4 or more cervical disc levels or an occipital-cervical fusion.
* Actively being treated by a medical provider for concussion
* Known severe spinal deformity requiring medical treatment (e.g. scoliosis)
* Has been diagnosed by a medical provider with severe vertigo, fainting, narcolepsy, or balance disorders with high risk for falling
* Any known fractures within the last 3 months that will interfere with the motion assessment
* Any known spine fractures within the last 6 months
* Known unstable spondylolisthesis (i.e. standing 3mm of movement on flexion/extension film)
* Current condition requiring immobilization of the spine
* History of brain or spine cancer
* Currently or within the last 90 days, been treated for any cancer with chemotherapy or radiation therapy
* Known severe osteoporosis requiring medical treatment and physician-recommended physical restrictions
* Current open wounds or medical device entry points where the harnesses will be placed on the neck or back
* Current osteomyelitis or spine infection
* Any other reason that a treating physician, researcher, or participant determines it is unsafe for a patient to perform test

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: There are 3 different study populations: Controls/Insincere, Low Back Pain, and Neck Pain
Sampling Method: Non-Probability Sample
Enrollment: 10500 (Estimated)
Dates: Start 2020-12-18 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Motion Index | 2030
  Composite functional score ranging from 0 - 100, with higher scores indicating healthier function. This is a composite metric derived from a standardized sensor-enabled spinal motion assessment. Motion features extracted from the motion assessment are benchmarked against a normative population.
Patient's Global Impression of Change (PGIC) | 2030
  PGIC is a 7 point scale indicating a patient's preception of overall improvement after treatment. Patients rate their change as "very much improved," "much improved," "minimally improved," "no change," "minimally worse," "much worse," or "very much worse."

SECONDARY OUTCOMES:
PROMIS-29 | 2030
  The PROMIS-29 captures data from 7 domains ranging from Pain intensity, Pain Interference, Physical Function, Depression, Anixety, Fatigue, Sleep Disturbance, and Social Role
Pain Catastrophizing scale (PCS-6) | 2030
  PCS is used to characterize pain catastrophizing behaviors. It ranges between 0 - 24, with higher scores indicating more catastrophizing tendencies

CONTACTS AND LOCATIONS:
Locations (1):
- The Ohio State University Wexner Medical Center, Columbus, Ohio, United States

REFERENCES:
- [Derived] Mageswaran P, Dufour J, Aurand A, Knapik G, Hani H, Blakaj DM, Khan S, Hussain N, Tiwari M, Vallabh J, Weaver T, Marras WS. Wearable motion-based platform for functional spine health assessment. Reg Anesth Pain Med. 2024 Jul 8;49(7):518-527. doi: 10.1136/rapm-2023-104840. PMID 37813527